CLINICAL TRIAL: NCT03820115
Title: Effect of Elastic Abdominal Binder on Pain and Functional Recovery After Open Abdominal Surgery for Benign Gynecologic Conditions: a Randomized Controlled Trial
Brief Title: Elastic Abdominal Binder After Open Abdominal Surgery for Benign Gynecologic Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Kittipat Charoenkwan, MD, Associate Professor, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OBG-2561-05421
Record Dates: First submitted 2019-01-25; First posted 2019-01-29 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Gynecologic Disease
MeSH Terms: conditions — Genital Diseases, Female

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elastic abdominal binder (Experimental)
  Interventions: Device: Elastic abdominal binder
- No binder (No Intervention)

INTERVENTIONS:
Device: Elastic abdominal binder — Each woman in the intervention group is fitted with an elastic abdominal binder at the time of procedure completion just before leaving the operating room. The binder is placed snuggly tight (keeping in mind patient's comfort) on top of the hospital gown with the incision positioned at the middle part of the binder. The patients are encouraged to wear binders at all time. However, periods of break from wearing the binder are allowed at their convenience.
  Arms: Elastic abdominal binder

SUMMARY:
Surgery remains the backbone of modern management of benign gynecologic conditions. Some common surgical procedures include hysterectomy for uterine leiomyoma or adenomyosis, adnexectomy for ovarian and tubal pathology, and other conservative surgeries. These procedures can be accomplished by different surgical approaches comprising abdominal, vaginal, and laparoscopic routes. Although the use of vaginal and laparoscopic approach has increased in recent years, the open abdominal route is still the most commonly employed approach. This is especially the case in developing countries where resources to support the more expensive approach such as laparoscopy are quite limited. However, the procedure can be associated with significant morbidity. Delayed functional recovery influenced by pain and immobilization are important contributing factors for increased morbidity. Elastic abdominal binder, a wide elastic belt that is wore around the patient's abdomen to support surgical incision after surgery, has been employed by clinicians for pain relief, wound complications prevention, improved pulmonary function, and stabilization. Benefits of the abdominal binder use in this patient population have not been properly examined.

The aim of this study is to examine the effect of postoperative elastic abdominal binder use on recovery by comparing pain scores and mobility function (through the 6-minute walk test [6MWT]) in postoperative gynecologic patients who use versus do not use the elastic abdominal binder to support incisional site.

ELIGIBILITY:
Inclusion Criteria:

* Women, diagnosed with benign gynecologic conditions, undergoing open abdominal surgery

Exclusion Criteria:

* Surgeries performed for cancer
* Intraoperative accidental injury to urinary or gastrointestinal organs
* Postoperative admission to intensive care unit (ICU)
* Postoperative intraperitoneal drain placement
* Unable to understand and follow oral/written instructions
* Severe neuromuscular or circulatory disorders

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2019-05-31 (Actual)

PRIMARY OUTCOMES:
Daily average postoperative pain scores | An average of pain scores at 8:00 am and 4:00 pm, up to 7 days postoperation
  The participants are asked to rate postoperative pain according to 10-cm visual analog scales from '0' (no pain) to '10' (worst possible pain).
Six-minute walk test score change from baseline | One day before operation and postoperative day 3
  Six-minute walk test (6MWT)

SECONDARY OUTCOMES:
Rate of postoperative complications | In the morning, up to 7 days postoperation
  The complications of interest include febrile morbidity, wound complication, bowel ileus

CONTACTS AND LOCATIONS:
Overall Officials: Kittipat Charoenkwan, MD, MSc, Principal Investigator — Chiang Mai University
Locations (1):
- Kittipat Charoenkwan, Chiang Mai, Thailand